CLINICAL TRIAL: NCT00282932
Title: A Randomized, Double Blind, Placebo Controlled Detrol LA "Add-On" To Alpha-Blocker Study In Men With Persistent Overactive Bladder Symptoms Of Urinary Frequency And Urgency With/Without Urgency Incontinence After Previous Monotherapy With Alpha Blocker.
Brief Title: Detrol LA In Men With Overactive Bladder.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6121127
Record Dates: First submitted 2006-01-26; First posted 2006-01-27 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Overactive Bladder (OAB)
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Tolterodine Tartrate

INTERVENTIONS:
Drug: Detrol LA

SUMMARY:
An interventional active/placebo double blinded parallel randomized controlled study in which at 12 weeks of treatment, the primary endpoint of patient perception of bladder condition is measured along with associated safety and other secondary endpoints like bladder diary endpoints, quality of life and patient treatment satisfaction.

Patients included in the study must have symptoms of OAB (frequency of at least 8 per day and Urgency of at least 1 episode per day confirmed by bladder diary).

Patients are not eligible to enroll in the study if they have/had significant hepatic or renal disease, history of radiation treatment.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of OAB (frequency more than 8 per day and Urgency more than 1 episode per day confirmed by bladder diary)

Exclusion Criteria:

* Significant hepatic or renal disease, history of radiation treatment

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2006-01; Primary Completion 2007-05-01 (Actual); Study Completion 2007-05-14 (Actual)

PRIMARY OUTCOMES:
Patient Perception of Bladder Condition at 12 weeks of treatment

SECONDARY OUTCOMES:
1)To evaluate the additional benefit of 'Add-On' tolterodine L-tartrate ER (Detrol LA?), vs. placebo, to alpha-blocker therapy in men with persistent OAB symptoms of urinary frequency and urgency with/without urgency incontinence: a)On OAB symptoms as
assessed by 5-day voiding bladder diaries including Urinary Sensation Scale, b)On symptoms as assessed by the International Prostate Symptom Score (IPSS), c)On patient perception of treatment benefit as assessed by the Patient Perception of Treatment
Benefit Questionnaire (PPTB) , d)On patient perception of bladder condition as assessed by the change in the PPBC after 4 weeks of treatment, e)On bothersome quality of life (QoL) symptoms as assessed by the Overactive Bladder Questionnaire (OAB-q),
f)On sexual QoL as assessed by the ICIQ-MLUTSsex Questionnaire , g)On patient satisfaction with medication as assessed by the Overactive Bladder Treatment Satisfaction Questionnaires (OAB-s), h)On nocturia bothersome measure as assessed by the Nocturia
Quality-of-Life Questionnaire, 2)To evaluate the safety and tolerability of 'Add-On' tolterodine L-tartrate ER (Detrol LA?), vs. placebo, to alpha-blocker therapy in men with persistent OAB symptoms of urinary frequency and urgency with/without urgency
incontinence.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (72):
- United States (11):
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, La Mesa, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Iowa City, Iowa
  - Pfizer Investigational Site, Shreveport, Louisiana
  - Pfizer Investigational Site, Watertown, Massachusetts
  - Pfizer Investigational Site, Woodlane, New Jersey
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, State College, Pennsylvania
  - Pfizer Investigational Site, Houston, Texas
- Canada (9):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Surrey, British Columbia
  - Pfizer Investigational Site, Victoria, British Columbia
  - Pfizer Investigational Site, Kingston, Ontario
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Oakville, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Pointe-Claire, Quebec
- Denmark (3):
  - Pfizer Investigational Site, Aalborg
  - Pfizer Investigational Site, Herlev
  - Pfizer Investigational Site, Nykøbing Falster
- Germany (7):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Duisburg
  - Pfizer Investigational Site, Frankfurt
  - Pfizer Investigational Site, Muelheim A.d. Ruhr
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Rosenheim
  - Pfizer Investigational Site, Starnberg
- Italy (2):
  - Pfizer Investigational Site, Latina
  - Pfizer Investigational Site, Padua
- Mexico (4):
  - Pfizer Investigational Site, Guadalajara, Jalisco
  - Pfizer Investigational Site, Zapopan, Jalisco
  - Pfizer Investigational Site, Tlalpan, México DF
  - Pfizer Investigational Site, Durango
- Norway (2):
  - Pfizer Investigational Site, Bodø
  - Pfizer Investigational Site, Moelv
- Slovakia (5):
  - Pfizer Investigational Site, Bratislava
  - Pfizer Investigational Site, Košice
  - Pfizer Investigational Site, Malacky
  - Pfizer Investigational Site, Martin
  - Pfizer Investigational Site, Skalica
- South Africa (5):
  - Pfizer Investigational Site, Bloemfontein, Free State
  - Pfizer Investigational Site, Parktown, Gauteng
  - Pfizer Investigational Site, Durban, KwaZulu-Natal
  - Pfizer Investigational Site, Pietermaritzburg, KwaZulu-Natal
  - Pfizer Investigational Site, Cape Town
- South Korea (3):
  - Pfizer Investigational Site, Bucheon-si, Gyunggi-do
  - Pfizer Investigational Site, Busan
  - Pfizer Investigational Site, Seoul
- Spain (6):
  - Pfizer Investigational Site, A Coruña, A Coruña
  - Pfizer Investigational Site, Palma de Mallorca, Balearic Islands
  - Pfizer Investigational Site, Barcelona
  - Pfizer Investigational Site, Granada
  - Pfizer Investigational Site, Madrid
  - Pfizer Investigational Site, Valencia
- Sweden (4):
  - Pfizer Investigational Site, Borås
  - Pfizer Investigational Site, Huskvarna
  - Pfizer Investigational Site, Lund
  - Pfizer Investigational Site, Skövde
- Taiwan (3):
  - Pfizer Investigational Site, Hualien City
  - Pfizer Investigational Site, Kaohsiung City
  - Pfizer Investigational Site, Taipei
- Turkey (Türkiye) (4):
  - Pfizer Investigational Site, Adana
  - Pfizer Investigational Site, Istanbul
  - Pfizer Investigational Site, Izmir
  - Pfizer Investigational Site, Sihhiye-Ankara
- United Kingdom (4):
  - Pfizer Investigational Site, Bristol, Avon
  - Pfizer Investigational Site, Crewe, Cheshire
  - Pfizer Investigational Site, Taunton, Somerset
  - Pfizer Investigational Site, London

REFERENCES:
- [Derived] Chapple C, Herschorn S, Abrams P, Sun F, Brodsky M, Guan Z. Tolterodine treatment improves storage symptoms suggestive of overactive bladder in men treated with alpha-blockers. Eur Urol. 2009 Sep;56(3):534-41. doi: 10.1016/j.eururo.2008.11.026. Epub 2008 Nov 24. PMID 19070418
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6121127&StudyName=Detrol%20LA%20In%20Men%20With%20Overactive%20Bladder.%0D